CLINICAL TRIAL: NCT01481701
Title: A Non Randomized Stratified Phase II Trial Evaluating Efficacy and Safety of Oxaliplatin in Combination With 5-Fluorouracil in Patients With Platinum-sensitive and Platinum-resistant Recurrent Ovarian Carcinoma
Brief Title: A Trial Evaluating Efficacy and Safety of Oxaliplatin With 5-Fluorouracil in Patients With Recurrent Ovarian Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Folfox
Record Dates: First submitted 2011-07-18; First posted 2011-11-29 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2013-09

CONDITIONS: Ovarian Carcinoma; Relapse
Keywords: ovarian carcinoma; Bordet; relapse
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intravenous chemotherapy (Experimental): treatment of ovarian carcinoma in relapse
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — 85 mg/m² / 14days
  Other Names: No other intervention
Drug: oxaliplatin — oxaliplatin

SUMMARY:
This is a Phase II study for recurrent ovarian carcinoma platinum-sensitive and resistant tumors Folfox regimen.

DETAILED DESCRIPTION:
Evaluation of the safety and the efficacy of a combination of oxaliplatin and 5FU (Folfox) in patients with ovarian carcinoma relapsing either after platinum-combined regimen.

The Folfox regimen is administered every 14 days. Evaluation of the toxicity is performed at each cycle and evaluation of the efficacy every 4 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ovarian carcinoma relapse

Exclusion Criteria:

* neurotoxicity grade III renal clearance < 60 ml/min

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate | at 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Veronique D'Hondt, MD,PhD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium